CLINICAL TRIAL: NCT02345590
Title: Eplerenone in the Management of Abdominal Aortic Aneurysms: A Proof-Of-Concept Randomised Controlled Trial
Brief Title: Eplerenone in the Management of Abdominal Aortic Aneurysms
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01/15
Record Dates: First submitted 2015-01-11; First posted 2015-01-26 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eplerenone (Experimental): 25mg Eplerenone once daily for 12 months
  Interventions: Drug: Eplerenone
- Matching placebo (Placebo Comparator): Matching placebo once daily for 12 months
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — 25mg of eplerenone
  Other Names: Inspra

SUMMARY:
Weakening and expansion of the main abdominal artery (abdominal aortic aneurysm, AAA) is a common problem in older Australians. The majority of AAAs are small (<55 mm) and affect 90,000 individuals in Australia and 4.5 million world-wide. Currently, the only treatment available for AAA is surgery. However, surgical therapies are not effective for small AAAs, and these patients undergo a program of repeat imaging and consultation to monitor the size of the aneurysm and symptoms.

This proposal is aimed at addressing the urgent need to identify a medical treatment able to limit progression of AAAs.

The study design and rationale are based on strong preclinical evidence supporting the value of eplerenone (an agent indicated for treatment of heart failure) in limiting AAA progression. If proved effective, this medication would:

1. Reduce the number of patients requiring costly surgery
2. Reduce the number of surgery related deaths and complications
3. Provide a therapy suitable for the rapidly expanding elderly age group who have AAAs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged over 60years (inclusive); AAA measuring a maximum diameter of 30-49 mm on MRI; no current indication for AAA repair according to the treating physician or expectation that this will be revised within the next year; high likelihood of compliance with treatment over 12 months; stable medication regime for the last six months; have given signed informed consent to participate in the study.

Exclusion Criteria:

* Serum potassium concentration of more than 5.0 mmol/L before randomisation; evidence of renal impairment defined as serum creatinine>133 umol/L or creatinine clearance of <60 mL/min; known significant renal stenosis (>70%) of one or both renal arteries; evidence of liver disease (i.e. cirrhosis or hepatitis) or abnormal liver function defined as aspartate aminotransferase, alanine aminotransferase or total bilirubin >1.5x the upper limit of normal; evidence of primary aldosteronism (plasma aldosterone/renin ratio>650 pmol/L); electrolyte imbalance; active gout; use of MR antagonists; use of potassium-sparing diuretics, or potassium supplements; individuals with claustrophobia or a history of any metallic prosthetic implant contraindicating MRI.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
abdominal aortic aneurysm maximum orthogonal diameter | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Leah Isles, MBBS, Principal Investigator — The Alfred
Locations (2):
- Australia (2):
  - Baker IDI, Melbourne, Victoria
  - Heart Centre, Alfred Health, Melbourne, Victoria